CLINICAL TRIAL: NCT01583101
Title: Increasing Prompt Response Rates in the CHICA System
Brief Title: Child Health Improvement Through Computer Automation (CHICA) Highlighting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Aaron Carroll, Assoc. Prof of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHICA_Highlight_Study
Record Dates: First submitted 2012-04-18; First posted 2012-04-23 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Physician Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receiving Highlighted Prompts (Experimental): Prompts received by physicians were highlighted.
  Interventions: Other: Receiving Highlighted Prompts
- Receiving Non-highlighted Prompts (Active Comparator): Prompts received by physicians were not highlighted.
  Interventions: Other: Receiving Non-highlighted Prompts

INTERVENTIONS:
Other: Receiving Highlighted Prompts — Prompts received by physicians were highlighted.
  Arms: Receiving Highlighted Prompts
Other: Receiving Non-highlighted Prompts — Prompts received by physicians were not highlighted.
  Arms: Receiving Non-highlighted Prompts

SUMMARY:
The investigators have developed a novel decision support system for implementing clinical guidelines in pediatric practice. CHICA (Child Health Improvement through Computer Automation) combines three elements: (1) pediatric guidelines encoded in Arden Syntax; (2) a dynamic, scannable paper user interface; and (3) an HL7-compliant interface to existing electronic medical record systems. The result is a system that both delivers "just-in-time" patient-relevant guidelines to physicians during the clinical encounter, and accurately captures structured data from all who interact with it. Preliminary work with CHICA has demonstrated the feasibility of using the system to implement and evaluate clinical guidelines.

However, analyses have shown that physicians ignore a fair number of prompts. The investigators would like to experiment with changes to the system to see if they can increase physicians' response rates. This could include highlighting prompts, reordering them, or flagging them in other ways. The main outcome of interest in the rate at which physicians answer prompts.

DETAILED DESCRIPTION:
We have developed a novel decision support system for implementing clinical guidelines in pediatric practice. CHICA (Child Health Improvement through Computer Automation) combines three elements: (1) pediatric guidelines encoded in Arden Syntax; (2) a dynamic, scannable paper user interface; and (3) an HL7-compliant interface to existing electronic medical record systems. The result is a system that both delivers "just-in-time" patient-relevant guidelines to physicians during the clinical encounter, and accurately captures structured data from all who interact with it. Preliminary work with CHICA has demonstrated the feasibility of using the system to implement and evaluate clinical guidelines.

However, analyses have shown that physicians ignore a fair number of prompts. We would like to experiment with changes to the system to see if we can increase physicians' response rates. This could include highlighting prompts, reordering them, or flagging them in other ways. The main outcome of interest is the rate at which physicians answer prompts.

This will be a randomized, controlled trial of the CHICA system to see if we can improve prompt response rates. We will randomize physicians or clinics to receive some form of prompt change, including highlighting them, reordering them, or flagging them. No other changes will be made to care.

We will extract data from the CHICA system for all patients seen in our study clinics. This data will include a the clinic location, whether or not a physician responded to a prompt, the prompt's position on the form, the patient's gender, the rule priority of the prompt, rule title, patient insurance category, the patient's age in days, and the name of the provider. The main outcome of interest is whether or not a prompt was answered (discussed/not discussed).

ELIGIBILITY:
Inclusion Criteria:

* Physicians practicing in one of our four CHICA clinics who use CHICA

Exclusion Criteria:

* Not being a physician practicing in one of our four CHICA clinics who use CHICA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2237 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IUMG Clinic System, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While physicians were the ones that received prompts, the prompts are the unit of analysis.
Groups:
- Highlighted Prompts: Physicians received highlighted prompts.
- Non-highlighted Prompts: Physicians received prompts that were not highlighted.
Period: Overall Study
Arm/Group | Highlighted Prompts | Non-highlighted Prompts
Started | 1076 | 1161
Completed | 1076 | 1161
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Receiving Highlighted Prompts: These patients received highlighted prompts.
- Receiving Non-highlighted Prompts: These patients received prompts that were not highlighted.
- Total: Total of all reporting groups
Arm/Group | Receiving Highlighted Prompts | Receiving Non-highlighted Prompts | Total
Number analyzed (Participants) | 1076 | 1161 | 2237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1076 | 1161 | 2237
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — We did not record gender for this study, and so it is not known.
  Participants
    Unknown | 1076 | 1161 | 2237

OUTCOME MEASURES:

1. Primary Outcome: The Number of Prompts That Were Responded to
Description: The main outcome of interest is whether or not a prompt was answered (discussed/not discussed).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Receiving Highlighted Prompts | Receiving Non-highlighted Prompts
Number analyzed (Participants) | 1076 | 1161
Participants | 672 | 712

ADVERSE EVENTS:
Groups:
- Highlighted Prompts: These patients received highlighted prompts.
- Non-highlighted Prompts: These patients received prompts that were not highlighted.
Arm/Group | Highlighted Prompts | Non-highlighted Prompts
Serious Adverse Events (participants affected / at risk) | 0/1076 | 0/1161
Other Adverse Events (participants affected / at risk) | 0/1076 | 0/1161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No